CLINICAL TRIAL: NCT01834131
Title: Comprehensive Approach for Hypertension Prevention and Control in Argentina
Brief Title: Hypertension Control Program in Argentina (HCPIA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Institute for Clinical Effectiveness and Health Policy (Other)
Responsible Party: Principal Investigator, Jiang He, MD, PhD, Professor and Chair, Department of Epidemiology, Tulane University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U01HL114197 (NIH); U01HL114197 (NIH)
Record Dates: First submitted 2013-04-13; First posted 2013-04-17 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Hypertension
Keywords: hypertension; community health worker; home health education; medication adherence; mobile health; physician education; home blood pressure monitoring; implementation
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Clinics assigned to usual care will not receive any of the intervention components. Physicians in these clinics will continue to treat patients using their usual methods. Participants from these clinics will not receive community health worker visits or the mobile health intervention
- Comprehensive Intervention (Experimental): 1. Physicians will receive training in the use of treatment algorithms based on hypertension guidelines.
  2. Community health workers (CHW) will be trained in facilitating behavioral change through BP monitoring, medication management, and lifestyle modifications. CHW will serve as a source of education, motivation, and social support, and as facilitators of healthcare utilization for participants. CHW will conduct home visits, schedule appointments with primary care physicians, deliver antihypertensive medications to patients' homes, and provide tailored counseling to address barriers to behavior change.
  3. Individualized text messages to promote lifestyle changes and reminders to reinforce medication adherence will be sent to participants weekly.
  Interventions: Behavioral: Comprehensive Intervention

INTERVENTIONS:
Behavioral: Comprehensive Intervention — The comprehensive intervention includes physician education, a community health worker home intervention and a mobile health intervention. Please see Arm Description for details.
  Arms: Comprehensive Intervention

SUMMARY:
The objective of this cluster randomized trial is to test whether a comprehensive intervention program within a national public primary care system will improve hypertension control among uninsured hypertensive patients and their families in Argentina.

DETAILED DESCRIPTION:
Background: Although the efficacy and effectiveness of lifestyle modifications and antihypertensive pharmaceutical treatment for the prevention and control of hypertension and concomitant cardiovascular disease and premature death have been demonstrated in randomized controlled trials, this scientific knowledge has not been fully applied in the general population, especially in low and middle income countries.

Objectives: To test whether a comprehensive intervention program within a national public primary care system will improve hypertension control among uninsured hypertensive patients and their families in Argentina

Design: Cluster randomized trial

Study Participants: 1,890 study participants from 18 primary care clinics within a public primary care network in Argentina will be recruited. Patients with hypertension from the participating clinics, their spouses, and their adult hypertensive family members will be enrolled.

Intervention: Nine clinics with approximately 945 participants will be randomly assigned to the comprehensive intervention group and 9 clinics with similar participants to the usual care group. The comprehensive intervention, including health care provider education, a home-based intervention among patients and their families (lifestyle modification and home blood pressure [BP] monitoring) delivered by community health workers, and a mobile health intervention, will last for 18 months.

Outcomes: BP and other indicators will be measured at baseline and months 6, 12, and 18 during follow-up using standard methods. The primary outcome is a net change in systolic (SBP) and diastolic BP (DBP) from baseline to month 18 between the intervention and control groups among hypertensive study participants. The secondary outcomes are the proportion of hypertensive patients with adequate BP control (BP<140/90 mmHg), cost-effectiveness of hypertension control, and net BP changes in normotensive participants.

ELIGIBILITY:
Inclusion Criteria for Clinics:

* The clinic is affiliated with the Remediar+Redes program.
* The clinic is located in urban poor areas according to the 2010 census data.
* The clinic has ≥1000 outpatient visits each month, so that sufficient participants can be recruited.
* The minimum distance between the selected clinics will be 10 kilometers to minimize the risk for contamination of the intervention.
* Physician visits and essential medications are free of charge to patients under all circumstances.
* The clinic has a high number of prescriptions for antihypertensive medications.
* The clinic employs community health workers.
* The clinic has general practitioners and nurses.
* The clinic has a history of good performance in the Remediar+Redes program.
* The clinic performs blood draws on patients when appropriate.

Inclusion Criteria for Participants:

* Patients aged ≥21 years who received primary care from the participating clinics and have hypertension ( SBP ≥140 mmHg and/or DBP ≥90 mmHg on at least 2 separate visits) and their spouses (with or without hypertension) and/or any adult hypertensive family members (age ≥21 years) living in the same household will be included.
* Hypertension patients and their spouses and/or family members must be available for the first baseline nurse home visit.
* The index patient must have a cell phone that receives text messages.
* The family's homes must be located within 10 kilometers from the clinic.

Exclusion Criteria for Participants:

* Hypertension patients who do not have a spouse or another adult with hypertension in the household.
* Plans to move from the neighborhood in the next two years
* Pregnant women or women who are planning to become pregnant in the next two years
* Persons who are bed-bound
* Persons who cannot give informed consent
* Persons with an arm circumference >50 cm

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1954 (Actual)
Dates: Start 2013-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Net change in systolic (SBP) and diastolic BP (DBP) from baseline to month 18 between the intervention and control groups among hypertensive study participants. | Baseline and 18 months
  Three BP measurements will be obtained at each data collection visit by study nurses who are masked to clinic assignment. BP will be measured according to a standard protocol recommended by the American Heart Association. The average of the three measurements will be used to compare the change over 18 months between the intervention and control groups.

SECONDARY OUTCOMES:
Proportion of hypertension control (BP<140/90 mmHg) among hypertensive patients | Baseline and 18 months
  The proportion of hypertensives with blood pressure control (defined as (BP<140/90 mmHg or < 130/80 mmHg if patient has diabetes of CKD) will be compared between the intervention and control group.
Self-reported medication adherence among hypertensive patients | Baseline and 18 months
  The Morisky scale questionnaire will be administered at baseline and 18 months of follow-up to compare medication adherence between the intervention and control groups.
Cost-effectiveness of the intervention | Baseline and 18 Months
  All resources involved in conducting this comprehensive intervention program, as well as all patient-level costs, will be documented. Primary incremental cost effectiveness ratio (ICER) measure will be cost per mmHg of change in SBP and DBP.
Net change in systolic (SBP) and diastolic BP (DBP) from baseline to month 18 between the intervention and control groups among normotensive study participants | Baseline and 18 months
  Three BP measurements will be obtained at each data collection visit by study nurses who are masked to clinic assignment. BP will be measured according to a standard protocol recommended by the American Heart Association. The average of the three measurements will be used to compare the change over 18 months between the intervention and control groups among normotensives.
Net change in body weight and waist circumference from baseline to 18 months | Baseline and 18 months
  Study nurses will take anthropometric measurements on individuals in light clothing without shoes using a standard protocol.
Intensity of treatment | Baseline and 18 months
  Intensification (titration and/or addition) of antihypertensive medications,compared between the intervention and control groups after 18 months of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang He, MD, PhD, Principal Investigator — Tulane University Health Sciences Center
Locations (1):
- Institute for Clinical Effectiveness and Health Policy, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
Our study data sharing plan will comply with all NIH policies for data sharing. Sharing of data and scientific findings with the research and clinical communities will be executed through the centralized NIH data repository, publications in peer reviewed journals, and presentations at scientific meetings. Data sharing will be implemented in a timely manner. The study data, including data from baseline and follow-up visits, will be prepared for transmission to the NHLBI data repository beginning two years after the last subject completes the study visit. These data will be free of identifiers that allow identification of individual research participants either directly or through "deductive disclosure." In addition, we will offer through our public access website opportunities for outside investigators to collaborate with us using the complete study data and samples.
Supporting Information: Study Protocol
Time Frame: Immediately after main paper published.

REFERENCES:
- [Background] Mills KT, Bundy JD, Kelly TN, Reed JE, Kearney PM, Reynolds K, Chen J, He J. Global Disparities of Hypertension Prevalence and Control: A Systematic Analysis of Population-Based Studies From 90 Countries. Circulation. 2016 Aug 9;134(6):441-50. doi: 10.1161/CIRCULATIONAHA.115.018912. PMID 27502908
- [Result] Mills KT, Rubinstein A, Irazola V, Chen J, Beratarrechea A, Poggio R, Dolan J, Augustovski F, Shi L, Krousel-Wood M, Bazzano LA, He J. Comprehensive approach for hypertension control in low-income populations: rationale and study design for the hypertension control program in Argentina. Am J Med Sci. 2014 Aug;348(2):139-45. doi: 10.1097/MAJ.0000000000000298. PMID 24978148
- [Derived] Palmer MJ, Machiyama K, Woodd S, Gubijev A, Barnard S, Russell S, Perel P, Free C. Mobile phone-based interventions for improving adherence to medication prescribed for the primary prevention of cardiovascular disease in adults. Cochrane Database Syst Rev. 2021 Mar 26;3(3):CD012675. doi: 10.1002/14651858.CD012675.pub3. PMID 33769555
- [Derived] Poggio R, Melendi SE, Beratarrechea A, Gibbons L, Mills KT, Chen CS, Nejamis A, Gulayin P, Santero M, Chen J, Rubinstein A, He J, Irazola V. Cluster Randomized Trial for Hypertension Control: Effect on Lifestyles and Body Weight. Am J Prev Med. 2019 Oct;57(4):438-446. doi: 10.1016/j.amepre.2019.05.011. Epub 2019 Aug 29. PMID 31473065
- [Derived] He J, Irazola V, Mills KT, Poggio R, Beratarrechea A, Dolan J, Chen CS, Gibbons L, Krousel-Wood M, Bazzano LA, Nejamis A, Gulayin P, Santero M, Augustovski F, Chen J, Rubinstein A; HCPIA Investigators. Effect of a Community Health Worker-Led Multicomponent Intervention on Blood Pressure Control in Low-Income Patients in Argentina: A Randomized Clinical Trial. JAMA. 2017 Sep 19;318(11):1016-1025. doi: 10.1001/jama.2017.11358. PMID 28975305